CLINICAL TRIAL: NCT01189201
Title: Relative Bioavailability Investigations of a 25 mg BI 10773 / 5 mg Linagliptin Fixed Dose Combination (FDC) Tablet (Formulation A1) Including the Comparison With Its Mono-components, the Comparison With a Second FDC Tablet (Formulation A3), and the Investigation of Food (an Open-label, Randomised, Single Dose, Crossover, Phase I Trial in Healthy Male and Female Volunteers)
Brief Title: Rel. BA of Empagliflozin (BI 10773)/Linagliptin FDC Tbl, Comparison With Mono-components, With a Second FDC Tablet and Influence of Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1275.3; 2010-019211-38 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Linagliptin

ARMS (4):
- BI 10773/linagliptin FDC SID (Experimental): medium single dose ofBI 10773/linagliptin FDC (Formulation A1)
  Interventions: Drug: BI 10773/linagliptin
- BI 10773/linagliptin SID (Experimental): medium single dose of mono components BI 10773/linagliptin
  Interventions: Drug: BI 10773/linagliptin SID
- BI 10773/linagliptin FDC (Experimental): medium single dose of BI 10773/linagliptin FDC (Formulation A1) after high fat, high caloric meal
  Interventions: Drug: BI 10773/linagliptin FDC
- BI 10773/linagliptin (Experimental): medium single dose of BI 10773/linagliptin FDC (Formulation A3)
  Interventions: Drug: BI 10773/linagliptin

INTERVENTIONS:
Drug: BI 10773/linagliptin — medium single dose of BI 10773/linagliptin FDC (Formulation A1)
  Arms: BI 10773/linagliptin FDC SID
Drug: BI 10773/linagliptin — medium single dose of BI 10773/linagliptin FDC (Formulation A3)
  Arms: BI 10773/linagliptin
Drug: BI 10773/linagliptin SID — medium single dose of mono components BI 10773/linagliptin
  Arms: BI 10773/linagliptin SID
Drug: BI 10773/linagliptin FDC — medium single dose of BI 10773/linagliptin FDC (Formulation A1) after high fat, high caloric meal
  Arms: BI 10773/linagliptin FDC

SUMMARY:
The primary objective of the current study is to investigate the relative bioavailability of BI 10773 / linagliptin fixed dose combination tablet (formulation A1, Treatment A, Test) compared to BI 10773 given in free combination with linagliptin (Treatment B, Reference), both in the fasting state. All 42 subjects entered are planned to be included in this comparison.

The secondary objective is to investigate the relative bioavailability of BI 10773 / linagliptin fixed dose combination tablet after administration of a standardised high fat, high caloric meal (formulation A1, Treatment C, Test) compared to BI 10773 / linagliptin fixed dose combination in the fasting state (formulation A1,Treatment A, Reference). Of the 42 subjects entered 18 subjects are planned to be included in this comparison.

An additional objective is to investigate the relative bioavailability of a second formulation of the fixed dose combination tablet of BI 10773 / linagliptin (formulation A3,Treatment D, Test) compared to BI 10773 / linagliptin fixed dose combination tablet (formulation A1,Treatment A, Reference). Of the 42 subjects entered 24 subjects are planned to be included in this comparison.

ELIGIBILITY:
Inclusion criteria:

healthy male and female subjects

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1275.3.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

REFERENCES:
- [Derived] Glund S, Mattheus M, Runge F, Rose P, Friedrich C. Relative bioavailability of an empagliflozin 25-mg/linagliptin 5-mg fixed-dose combination tablet . Int J Clin Pharmacol Ther. 2017 Apr;55(4):355-367. doi: 10.5414/CP202929. PMID 28290274

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Overall: A randomised, open label, three period, crossover trial. Each subject was to receive 3 of 4 possible treatments. The treatments were
  * Empagliflozin plus linagliptin fixed dose combination (FDC) A1 (fasted)
  * Empagliflozin plus linagliptin, individual tablets (fasted)
  * Empagliflozin plus linagliptin FDC A1 (fed)
  * Empagliflozin plus linagliptin FDC A3 (fasted)
  Drug administrations were separated by a washout period of at least 35 days.
  A total of 42 subjects were entered into the study, all subjects were allocated to the FDC A1 (fasted) and individual tablet treatments as this was the primary objective of the study. Along with this 18 of the subjects were allocated to receive the FDC A1 (fed) treatment and other 24 subjects to the FDC A3 treatment.
Period: Overall Study
Arm/Group | Study Overall
Started | 42
Received Empa/Linagliptin FDC A1(Fasted) | 42
Rec. Empa/Linagliptin Ind.Tablet(Fasted) | 41
Received Empa/Linagliptin FDC A1 (Fed) | 18
Received Empa/Linagliptin FDC A3(Fasted) | 24
Completed | 41
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Study Overall
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Empagliflozin: Area Under the Curve 0 to the Last Quantifiable Drug Plasma Concentration (AUC0-tz)
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma over the time interval from 0 to the last quantifiable drug plasma concentration.
  In this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: 1 hour (h) before drug administration and 20 minutes (min), 40min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h, 72h after drug administration
Population: Pharmacokinetic (PK) set: Included all subjects who were documented to have taken at least one dose of investigational treatment, who provided at least one observation for at least one primary endpoint without important protocol violations relevant to the PK evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Empa Plus Linagliptin FDC A1 (Fasted): A single dose of empa 25 mg and linagliptin 5 mg fixed dose combination (FDC) tablet formulation A1 (FDC A1)
- Empa Plus Linagliptin Individual Tablets (Fasted): Individual tablets of empa 25 mg and linagliptin 5 mg administered together
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin Individual Tablets (Fasted)
Number analyzed (Participants) | 42 | 40
nmol*h/L | 5990 (21.0) | 5720 (20.8)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin Individual Tablets (Fasted); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin individual tablets (fasted); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 104.90, 90% CI 2-sided [102.07 to 107.80], Standard Deviation 7.2 — Standard deviation is actually the geometric coefficient of variation (gCV)

2. Primary Outcome: Linagliptin: Area Under the Curve 0 to 72 Hours (AUC0-72)
Description: Area under the concentration-time curve of linagliptin in plasma over the time interval from 0 to 72 hours.
  In this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin Individual Tablets (Fasted)
Number analyzed (Participants) | 42 | 40
nmol*h/L | 264 (22.1) | 250 (22.1)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin Individual Tablets (Fasted); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin individual tablets (fasted); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 104.91, 90% CI 2-sided [99.97 to 110.09], Standard Deviation 12.8 — Standard deviation is actually the gCV

3. Primary Outcome: Empagliflozin: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of empagliflozin (empa) in plasma.
  In this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin Individual Tablets (Fasted)
Number analyzed (Participants) | 42 | 40
nmol/L | 862 (26.8) | 803 (24.9)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin Individual Tablets (Fasted); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin individual tablets (fasted); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 107.68, 90% CI 2-sided [101.70 to 114.02], Standard Deviation 15.3 — Standard deviation is actually the gCV

4. Primary Outcome: Linagliptin: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of linagliptin in plasma.
  In this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin Individual Tablets (Fasted)
Number analyzed (Participants) | 42 | 40
nmol/L | 8.19 (36.4) | 7.49 (31.0)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin Individual Tablets (Fasted); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin individual tablets (fasted); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 109.68, 90% CI 2-sided [99.55 to 120.83], Standard Deviation 26.2 — Standard deviation is actually the gCV

5. Secondary Outcome: Empagliflozin: Time From Last Dosing to Maximum Measured Concentration (Tmax)
Description: Time from last dosing to the maximum measured concentration of empagliflozin (empa) in plasma.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Groups:
- Empa Plus Linagliptin FDC A1 (Fed): A single dose of empa 25 mg and linagliptin 5 mg FDC A1 tablet given after a high-fat, high-caloric meal.
- Empa Plus Linagliptin FDC A3 (Fasted): A single dose of empa 25 mg and linagliptin 5 mg FDC tablet formulation A3.
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin Individual Tablets (Fasted) | Empa Plus Linagliptin FDC A1 (Fed) | Empa Plus Linagliptin FDC A3 (Fasted)
Number analyzed (Participants) | 42 | 40 | 18 | 24
hours | 1.50 [0.67 to 4.00] | 1.25 [0.67 to 3.98] | 2.00 [0.67 to 4.00] | 1.50 [0.67 to 3.00]

6. Secondary Outcome: Linagliptin: Time From Last Dosing to Maximum Measured Concentration (Tmax)
Description: Time from last dosing to the maximum measured concentration of linagliptin in plasma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin Individual Tablets (Fasted) | Empa Plus Linagliptin FDC A1 (Fed) | Empa Plus Linagliptin FDC A3 (Fasted)
Number analyzed (Participants) | 42 | 40 | 18 | 24
hours | 1.50 [0.33 to 6.03] | 1.75 [0.67 to 10.0] | 2.25 [1.00 to 4.00] | 1.50 [0.33 to 4.00]

7. Secondary Outcome: Empagliflozin: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma over the time interval from 0 extrapolated to infinity.
  In this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin Individual Tablets (Fasted)
Number analyzed (Participants) | 42 | 40
nmol*h/L | 6060 (20.7) | 5800 (20.9)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin Individual Tablets (Fasted); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin individual tablets (fasted); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 104.78, 90% CI 2-sided [102.02 to 107.61], Standard Deviation 7.1 — Standard deviation is actually the gCV

8. Secondary Outcome: Linagliptin: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of linagliptin in plasma over the time interval from 0 extrapolated to infinity.
  In this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin Individual Tablets (Fasted)
Number analyzed (Participants) | 42 | 40
nmol*h/L | 435 (26.5) | 410 (29.8)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin Individual Tablets (Fasted); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin individual tablets (fasted); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 104.64, 90% CI 2-sided [97.23 to 112.62], Standard Deviation 19.7 — Standard deviation is actually the gCV

9. Secondary Outcome: Empagliflozin Fed vs Fasted: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: as for outcome 7
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin FDC A1 (Fed)
Number analyzed (Participants) | 18 | 18
nmol*h/L | 6410 (16.0) | 5500 (16.8)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin FDC A1 (Fed); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin FDC A1 (fed); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 85.86, 90% CI 2-sided [81.33 to 90.64], Standard Deviation 9.3 — Standard deviation is actually the gCV

10. Primary Outcome: Empagliflozin Fed vs Fasted: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of empagliflozin (empa) in plasma, comparing fed with fasted.
  In this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin FDC A1 (Fed)
Number analyzed (Participants) | 18 | 18
nmol/L | 949 (23.7) | 583 (21.7)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin FDC A1 (Fed); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin FDC A1 (fed); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 61.41, 90% CI 2-sided [54.10 to 69.71], Standard Deviation 22.0 — Standard deviation is actually the gCV

11. Primary Outcome: Empagliflozin Fed vs Fasted: Area Under the Curve 0 to the Last Quantifiable Drug Plasma Concentration (AUC0-tz)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin FDC A1 (Fed)
Number analyzed (Participants) | 18 | 18
nmol*h/L | 6330 (16.4) | 5400 (16.3)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin FDC A1 (Fed); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin FDC A1 (fed); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 85.32, 90% CI 2-sided [80.77 to 90.14], Standard Deviation 9.4 — Standard deviation is actually the gCV

12. Secondary Outcome: Linagliptin Fed vs Fasted: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: as for outcome 8
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin FDC A1 (Fed)
Number analyzed (Participants) | 18 | 18
nmol*h/L | 453 (24.2) | 421 (19.0)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin FDC A1 (Fed); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin FDC A1 (fed); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 93.18, 90% CI 2-sided [85.07 to 102.05], Standard Deviation 15.7 — Standard deviation is actually the gCV

13. Primary Outcome: Linagliptin Fed vs Fasted: Maximum Measured Concentration (Cmax)
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin FDC A1 (Fed)
Number analyzed (Participants) | 18 | 18
nmol/L | 8.97 (40.0) | 6.14 (17.0)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin FDC A1 (Fed); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin FDC A1 (fed); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 68.48, 90% CI 2-sided [58.59 to 80.03], Standard Deviation 27.2 — Standard deviation is actually the gCV

14. Primary Outcome: Linagliptin Fed vs Fasted: Area Under the Curve 0 to 72 Hours (AUC0-72)
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin FDC A1 (Fed)
Number analyzed (Participants) | 18 | 18
nmol*h/L | 275 (21.7) | 250 (19.2)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin FDC A1 (Fed); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin FDC A1 (fed); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 90.95, 90% CI 2-sided [84.24 to 98.19], Standard Deviation 13.2 — Standard deviation is actually the gCV

15. Secondary Outcome: Empagliflozin Formulation Comparison: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: as for outcome 7
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Empa Plus Linagliptin FDC A3 (Fasted): A single dose of empa 25 mg and linagliptin 5 mg FDC tablet formulation A3 (FDC A3).
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin FDC A3 (Fasted)
Number analyzed (Participants) | 24 | 24
nmol*h/L | 5810 (23.1) | 5560 (20.8)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin FDC A3 (Fasted); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin FDC A3 (fasted); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 95.64, 90% CI 2-sided [91.19 to 100.30], Standard Deviation 9.6 — Standard deviation is actually the gCV

16. Primary Outcome: Empagliflozin Formulation Comparison: Maximum Measured Concentration (Cmax)
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin FDC A3 (Fasted)
Number analyzed (Participants) | 24 | 24
nmol/L | 802 (27.0) | 787 (25.2)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin FDC A3 (Fasted); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin FDC A3 (fasted); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 98.04, 90% CI 2-sided [91.95 to 104.53], Standard Deviation 13.0 — Standard deviation is actually the gCV

17. Primary Outcome: Empagliflozin Formulation Comparison: Area Under the Curve 0 to the Last Quantifiable Drug Plasma Concentration (AUC0-tz)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin FDC A3 (Fasted)
Number analyzed (Participants) | 24 | 24
nmol*h/L | 5740 (23.3) | 5490 (21.1)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin FDC A3 (Fasted); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin FDC A3 (fasted); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 95.69, 90% CI 2-sided [91.17 to 100.43], Standard Deviation 9.8 — Standard deviation is actually the gCV

18. Secondary Outcome: Linagliptin Formulation Comparison: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: as for outcome 8
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin FDC A3 (Fasted)
Number analyzed (Participants) | 24 | 24
nmol*h/L | 423 (28.3) | 393 (33.8)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin FDC A3 (Fasted); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin FDC A3 (fasted); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 92.98, 90% CI 2-sided [86.36 to 100.09], Standard Deviation 14.9 — Standard deviation is actually the gCV

19. Primary Outcome: Linagliptin Formulation Comparison: Maximum Measured Concentration (Cmax)
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin FDC A3 (Fasted)
Number analyzed (Participants) | 24 | 24
nmol/L | 7.65 (32.7) | 7.93 (33.5)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin FDC A3 (Fasted); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin FDC A3 (fasted); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 103.71, 90% CI 2-sided [92.93 to 115.74], Standard Deviation 22.4 — Standard deviation is actually the gCV

20. Primary Outcome: Linagliptin Formulation Comparison: Area Under the Curve 0 to 72 Hours (AUC0-72)
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin FDC A3 (Fasted)
Number analyzed (Participants) | 24 | 24
nmol*h/L | 256 (22.4) | 247 (26.3)
Statistical Analysis 1: Comparison: Empa Plus Linagliptin FDC A1 (Fasted) vs Empa Plus Linagliptin FDC A3 (Fasted); No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus linagliptin FDC A1 (fasted) divided by empa plus linagliptin FDC A3 (fasted); ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 96.36, 90% CI 2-sided [89.78 to 103.42], Standard Deviation 14.3 — Standard deviation is actually the gCV

21. Secondary Outcome: Clinically Relevant Abnormalities for Physical Examination, Vital Signs, ECG, Blood Chemistry and Assessment of Tolerability by the Investigator
Description: Clinically Relevant Abnormalities for Physical Examination, Vital Signs, ECG, Blood Chemistry and Assessment of Tolerability by the Investigator. New abnormal findings or worsening of baseline conditions were reported as Adverse Events. Time frame for adverse event was until the end-of-study examination.
Time Frame: Drug administration until next treatment period/end-of-study examination, up to 36 days
Population: Treated set (TS) included all subjects who were documented to have taken at least one dose of investigational treatment.
Measure: Number; unit: participants
Groups:
- Empa Plus Linagliptin Indivdual Tablets (Fasted): Individual tablets of empa 25 mg and linagliptin 5 mg administered together
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin Indivdual Tablets (Fasted) | Empa Plus Linagliptin FDC A1 (Fed) | Empa Plus Linagliptin FDC A3 (Fasted)
Number analyzed (Participants) | 42 | 41 | 18 | 24
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment period and following washout period, up to 36 days
Arm/Group | Empa Plus Linagliptin FDC A1 (Fasted) | Empa Plus Linagliptin Individual Tablets (Fasted) | Empa Plus Linagliptin FDC A1 (Fed) | Empa Plus Linagliptin FDC A3 (Fasted)
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41 | 0/18 | 0/24
Other Adverse Events (participants affected / at risk) | 8/42 | 5/41 | 6/18 | 4/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empa Plus Linagliptin FDC A1 (Fasted) (N=42) | Empa Plus Linagliptin Individual Tablets (Fasted) (N=41) | Empa Plus Linagliptin FDC A1 (Fed) (N=18) | Empa Plus Linagliptin FDC A3 (Fasted) (N=24)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 4 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.